CLINICAL TRIAL: NCT02567487
Title: Comparison of TAP Block With Two Different Doses of Levobupivacaine for Postoperative Pain Management in Pediatric Patients
Brief Title: TAP Block With Two Different Doses of Levobupivacaine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Emel Uyar, Doctor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 931893045140401
Record Dates: First submitted 2015-09-17; First posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Levobupivacaine high volume (Active Comparator): TAP block with levobupivacaine 0.25% of 0.5 ml/kg under general anesthesia
  Interventions: Drug: Levobupivacaine
- Group Levobupivacaine low volume (Active Comparator): TAP block with levobupivacaine 0.25% of 0.25 ml/kg under general anesthesia
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Transversus abdominis plane block with levobupivacaine
  Other Names: Chirocaine

SUMMARY:
The aim of the current study is to investigate the effects of two different doses of levobupivacaine in TAP (transversus abdominus plane) block for postoperative management. For this purpose we planned to include 50 children aged between 2 and 12 that will undergo unilateral inguinal surgery.

The doses that will be used in the study were within usual dose limits which is stated in prospectus of the study drug.

DETAILED DESCRIPTION:
Fifty children undergoing TAP block were randomly divided into two groups as levobupivacaine 0.25% 0.5 ml/kg and levobupivacaine 0.25% 0.25 ml/kg. Postoperative pain was evaluated with observational pain scale and modified pediatric objective pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers planned to undergo unilateral inguinal surgery under TAP (ilioinguinal and iliohypogastric block) and general anesthesia
* Aged between 2 and 12

Exclusion Criteria:

* Patients with coagulation dysfunction
* Patients with chronic pain
* Patients having infection at the site of intervention
* Patients with a history of allergy
* Patients having chronic diseases (hepatic dysfunction, renal failure)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
postoperative VAS score <4 at postoperative 24 hours | Postoperative first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Alkis, Study Director — Ankara University Medical Faculty